CLINICAL TRIAL: NCT06685900
Title: A Single-center, Randomized Controlled Pilot Trial to Evaluate Efficacy and Safety of Symptom Improvement by Digital Therapeutics to Manage Hypotension Symptoms
Brief Title: Efficacy and Safety of Symptom Improvement by Digital Therapeutics to Manage Hypotension Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1-2024-0028
Record Dates: First submitted 2024-10-06; First posted 2024-11-13 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant and Sub-investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention group (EIG) (Experimental): the trial group that begins treatment in the 3-week of the total 15-week study period
  Interventions: Device: digital therapeutics
- Late intervention group (LIG) (Experimental): the comparator group that begins treament in the 9-week of the total 15-week study period
  Interventions: Device: digital therapeutics

INTERVENTIONS:
Device: digital therapeutics — Early intervention group will undergo app usage training, disease education, blood pressure measurements, orthostatic blood pressure measurements, and postprandial blood pressure measurements up to the third week of participation. From the fourth week onward, for a duration of 12 weeks, non-pharmacological treatment education will be provided through a digital therapeutic, and blood pressure will be measured according to a specified schedule.
  Arms: Early intervention group (EIG)
Device: digital therapeutics — Late intervention group will undergo app usage training, disease education, blood pressure measurements, orthostatic blood pressure measurements, and postprandial blood pressure measurements up to the ninth week of participation. From the tenth week onward, for a duration of 6 weeks, non-pharmacological treatment education will be provided through a digital therapeutic, and blood pressure will be measured according to a specified schedule.
  Arms: Late intervention group (LIG)

SUMMARY:
This clinical trial is an exploratory study aimed at assessing the efficacy and safety of a digital therapeutic for managing symptoms of hypotension, with the goal of providing evidence for the design of future confirmatory clinical research.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 and older with symptoms suspected to be related to dizziness due to hypotension within the past year.
2. Individuals who are able to walk and can participate in the study using a smartphone, or for whom cooperation from a guardian is available.

Exclusion Criteria:

1. Individuals diagnosed with causes of dizziness other than hypotension, such as benign paroxysmal positional vertigo or stroke, within the past year.
2. Severe anemia (history of Hb < 8.0 g/dL within the last 3 months).
3. Individuals unable to use a smartphone (Android phone) or smartwatch.
4. Individuals with a life expectancy of less than 1 year due to diseases such as malignant tumors.
5. Individuals diagnosed with severe heart valve disease or severe heart failure with LVEF < 35% (based on the most recent examination).
6. Recent rapid and unintended weight loss (5% or more, or 5 kg or more, within the last 6 months).

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
The number of hypotension symptom events | within the first 6weeks after intervention
  The effectiveness of symptom improvement for hypotension was evaluated in the trial and control groups based on the frequency of hypotension symptoms over a 6-week period.

SECONDARY OUTCOMES:
Number of symptoms related to hypotension | over 15weeks
  Comparison of the frequency of symptoms suspected to be caused by hypotension before and after the intervention
Number of falling accident | over 15weeks
  To investigate whether regularly measuring blood pressure can help prevent falls.
Details for disease diagnosis and concomitant medications | over 15weeks
  To idenfity the correlation between hypotension and other causes and symptoms
The frequency of use of digital therapeutics | at 15weeks
  To identify how many times participants use digital therapeutics to measure blood pressure.
  Display the frequency of data input through digital therapeutics as the mean or median.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university college of medicine, Seoul, South Korea